CLINICAL TRIAL: NCT01820832
Title: Phase 4 Study of Oral Calcitriol for Reduction of Mild Proteinuria in Patients With CKD
Brief Title: Oral Calcitriol for Reduction of Mild Proteinuria in Patients With CKD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Jing Chen, Professor, PhD., MD, Renal Division, Huashan Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Calcitriol-MP-1
Record Dates: First submitted 2013-03-19; First posted 2013-03-29 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Chronic Kidney Disease; Proteinuria
Keywords: mild proteinuria; calcitriol; renal function; blood pressure
MeSH Terms: conditions — Renal Insufficiency, Chronic; Proteinuria | interventions — Calcitriol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Calcitriol (Experimental): General treatments (such as blood pressure control, lipid lowering, and so on) plus Calcitriol 0.5 ug/BIW for 24 weeks.
  Interventions: Drug: Calcitriol
- Control (No Intervention): General treatments.

INTERVENTIONS:
Drug: Calcitriol — Calcitriol 0.5 ug/BIW for 24 weeks.
  Other Names: 1, 25 - dihydroxy Cholecalciferol
  Arms: Calcitriol

SUMMARY:
The safety and efficacy of Caltriol on mild proteinuria (<1.0g/d) reduction in CKD patients.

DETAILED DESCRIPTION:
Proteinuria is not only a capital sign of kidney disease, but also a marker of chronic kidney disease (CKD) progression. Emerging evidence in patients with CKD show that vitamin D and its analogs can reduce proteinuria or albuminuria in the presence of angiotensin-converting enzyme inhibithion. While some of the studies reported that vitamin D receptor activation has been associated with increased serum creatinine and reduced estimated glomerular filtration rates. Therefore, the investigators plan to conduct a randomized clinical study to evaluate the efficacy and safety of Calcitriol in the treatment of mild proteinuria (<1.0g/d) CKD patients,which has no specific treatment at present.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-75 years
* clinical diagnosed and/or biopsy-confirmed primary glomerulonephritis
* proteinuria 0.15-1.0 g/d in 2 consecutive samples within 4 weeks despite ACE inhibitor (ACEI) or angiotensin receptor blocker (ARB) treatment for at least 1 year or ACEI/ARB withdrawal because of of drug intolerances (low blood pressure, cough, hyperkalemia) for at least 1 month
* estimated glomerular filtration rate (eGFR)>60ml/min/1/73m2
* corticosteroid and immunosuppressive agents withdrawal for at least 6 months
* normal blood pressure
* serum intact parathyroid hormone (iPTH) level >20pg/mL
* corrected serum calcium level < or = 2.55 mmol/L
* serum phosphorus level < or = 1.68 mmol/L
* 24 hours urinary calcium excretion level < or = 7.5 mmol
* not receive treatment of vitamin D or its analogue within 6 months
* willigness to give written consent and comply with the study protocol

Exclusion Criteria:

* history of sensitivity or allergy to calcitriol or other vitamin D analogs
* pregnancy, lactating women
* history of severe coexisting disease such as, but not limited to, chronic liver disease, myocardial infarction, cerebrovascular accident, malignant hypertension
* history of malignancy
* history of extraskeletal calcification, hyperuricemia, gout, kidney stone, gall stone, bone diseases
* patients receiving drugs contains of calcium
* patients receiving cimetidine, trimethoprim, or other drugs which can increase tubular creatinine reabsorption
* participation in any other trials within 1 month
* history of non-compliance

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-12 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
the percentage change of proteinuia | 24 weeks

SECONDARY OUTCOMES:
the proportion of patients achieving at least a 15% decrease in proteinuria | 24 weeks

OTHER OUTCOMES:
mean change of renal function (serum creatine, cystatin C, eGFR) | 24 weeks
blood pressure | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jing Chen, M.D. PhD, Principal Investigator — Division of Nephrology, Huashan Hospital, Fudan University
Locations (1):
- Huashan Hospital, Fudan University, Shanghai, Shanghai Municipality, China